CLINICAL TRIAL: NCT01964807
Title: Cardiovascular Assessment of the Effects of Tobacco and Nicotine Delivery Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P0052956; P50CA180890 (NIH); 136316 (Other: University of California, San Francisco)
Record Dates: First submitted 2013-10-04; First posted 2013-10-17 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Adverse Effect of Other Agents Primarily Affecting the Cardiovascular System, Initial Encounter
Keywords: Cardiovascular; tobacco; cigarettes; secondhand cigarette smoke; SHS; smokeless tobacco; chewing tobacco; snus; electronic cigarettes; vapor; particles; oxidative stress; flow-mediated dilation (FMD); FMD
MeSH Terms: conditions — Tobacco Use; Vaping | interventions — Tobacco Products; Nicotine; Electronic Nicotine Delivery Systems; Tobacco Smoke Pollution; Temperature; Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cigarette smokers (Experimental): Will smoke 1 cigarette, National Institute of Drug Abuse (NIDA) test type with 16.6 mg nicotine; 1 cigarette, NIDA test type with <0.45 mg nicotine; perform sham smoking by puffing on a drinking straw. Each intervention will last 10 minutes, and each will take place one time, on one of 3 study visits, in random order.
  Interventions: Other: Cigarette, NIDA test type with 16.6 mg nicotine; Other: Cigarette, NIDA test type with <0.45 mg nicotine; Other: Sham Smoking
- Nonsmokers (Experimental): Will undergo secondhand cigarette smoke (SHS) exposure and conditioned, filtered air exposure. Each intervention will last 180 minutes, and each will take place one time, on one of 2 study visits, in random order.
  Interventions: Other: Secondhand cigarette smoke (SHS); Other: Conditioned, filtered air
- Smokeless tobacco users (Experimental): Will use 1 pouch of commercially available moist oral snuff and will chew gum (sham moist snuff). Each intervention will last 30 minutes, and each will take place one time, on one of 2 study visits, in random order.
  Interventions: Other: Moist snuff; Other: Sham Moist Snuff
- e-cigarette users (Experimental): Will use one electronic cigarette with 18 mg/ml nicotine, one electronic cigarette with no nicotine, and will perform sham smoking by puffing on a drinking straw. Each intervention will last 10 minutes, and each will take place one time, on one of 3 study visits, in random order.
  Interventions: Other: Electronic cigarette with 18 mg/ml nicotine; Other: Electronic Cigarette with no nicotine; Other: Sham Smoking

INTERVENTIONS:
Other: Cigarette, NIDA test type with 16.6 mg nicotine — Smoke a single cigarette for up to 10 minutes
  Other Names: Cigarette
  Arms: Cigarette smokers
Other: Cigarette, NIDA test type with <0.45 mg nicotine — Smoke a single low-nicotine cigarette for up to 10 minutes
  Other Names: Cigarette
  Arms: Cigarette smokers
Other: Electronic cigarette with 18 mg/ml nicotine — Use electronic cigarette with 18 mg/ml nicotine for 30 minutes
  Arms: e-cigarette users
Other: Electronic Cigarette with no nicotine — Use electronic cigarette with no nicotine for 30 minutes
  Arms: e-cigarette users
Other: Moist snuff — Use moist snuff for 30 minutes
  Other Names: commercially available moist oral snuff
  Arms: Smokeless tobacco users
Other: Sham Smoking — Sham smoking or e-cigarette use consists of puffing on a drinking straw for 10 minutes
  Arms: Cigarette smokers; e-cigarette users
Other: Secondhand cigarette smoke (SHS) — 180-minute exposure to SHS generated by controlled dilution of smoke from machine-smoked cigarettes
  Other Names: Environmental Tobacco Smoke (ETS); ETS; SHS
  Arms: Nonsmokers
Other: Conditioned, filtered air — Exposure to conditioned, filtered air for 180 minutes
  Other Names: Clean, filtered, temperature and humidity controlled air; Negative control for SHS exposure
  Arms: Nonsmokers
Other: Sham Moist Snuff — Chew gum for 30 minutes
  Other Names: Chewing gum; Negative control for moist oral snuff use
  Arms: Smokeless tobacco users

SUMMARY:
The overarching goal of this project is to develop a panel of cardiovascular risk biomarkers that can detect differences in the cardiovascular safety of various tobacco products, whether conventional, new or emerging, in order to help the FDA with the task of regulating them. This will be achieved through 4 aims:

Aim 1: Determine the relative contributions of nicotine and combustion products to the cardiovascular risk of active cigarette smoking.

Aim 2: Determine which cardiovascular risk biomarkers are affected by exposure to secondhand smoke.

Aim 3: Determine the cardiovascular risk of smokeless tobacco use.

Aim 4: Determine the cardiovascular risk of electronic cigarettes and the respective contributions of nicotine and electronic cigarette vapor.

DETAILED DESCRIPTION:
Cigarette smoking is a major cause of cardiovascular disease (CVD).1 In contrast, the cardiovascular risks of other popular tobacco products (smokeless tobacco), new tobacco products ( e-cigarettes) and proposed products (reduced nicotine cigarettes) are not adequately understood. The FDA will need information about the cardiovascular safety of these products to inform their regulatory decisions. While long-term clinical outcome studies of the cardiovascular risks of these tobacco products would be optimal, they take too long to provide the data that the FDA needs now. Disturbances in the function of vascular endothelium (the lining of arteries, which plays an important role in regulating vascular function) and the activation of the autonomic nervous system, as well as increased inflammation, oxidative stress and propensity to thrombosis (clotting), are key mechanisms in the progression of CVD and validated biomarkers of CVD risk. These biomarkers form the basis for our model to assess the CVD risks of tobacco product use and secondhand smoke exposure. We will conduct controlled, short-term exposures of human subjects to test products that provide a wide range of nicotine, particle, and other cardiovascular toxin concentrations to determine how these components associated with tobacco use adversely affect cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* All Groups: Age 18-50
* Can tolerate withholding their medications for two weeks at a time
* Group 1: Active smokers
* Group 2: Nonsmokers
* Group 3: Active users of smokeless tobacco
* Group 4: Active users of electronic cigarettes
* Additional Inclusion Criteria for E-Cigarette Users:
* Currently use ofe-cigarettes > 5 times a day
* Has used e-cigarettes for >3 months
* Additional Inclusion Criteria for Active Smokers: Currently smoke >5 cigarettes per day ≥ 1 pack year

Exclusion Criteria:

* Exclusion Criteria for all subjects
* Physician diagnosis of:
* asthma
* heart disease
* hypertension
* dyslipidemia
* thyroid disease
* diabetes
* renal or liver impairment
* glaucoma.
* Unstable psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder)
* current use of more than two psychiatric medications
* Pregnancy or breastfeeding (by history)
* Alcohol, opiate, cocaine, amphetamine or methamphetamine dependence within the past 5 years
* BMI > 35 and < 18
* Current opiate, cocaine, amphetamine or methamphetamine use (by history or urine test)
* Occupational exposure to smoke, dusts and fumes
* Concurrent participation in another clinical trial
* Unable to communicate in English
* Additional Exclusion Criteria for Active Smokers:
* Unable to hold marijuana for 1 week prior to each study visit.
* Exhaled carbon monoxide (CO) <10 ppm at each visit
* Negative salivary cotinine test using a rapid-read, over the counter test with 30 ng/ml cutoff
* Additional Exclusion Criteria for Nonsmokers:
* More than 1 pack year smoking history
* Quit smoking < 5 years ago
* Ever a daily marijuana smoker
* Smoked anything within the last 3 months
* Additional Inclusion Criteria for Smokeless Tobacco Users:
* Use of moist oral snuff > 5 times a day
* Has used moist oral snuff for at least 0.5 years
* Additional Exclusion Criteria for Smokeless Tobacco Users:
* Current smoker
* Quit smoking < 0.5 years ago
* Additional Exclusion Criteria for E-Cigarette Users:
* Current use of other tobacco products
* Unable to hold marijuana for 1 week prior to each study visit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-11-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Flow-mediated Dilation of the Brachial Artery | up to 3 hours after use of tobacco product
  Vascular function as measured by Flow-mediated Dilation of the Brachial Artery

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | up to 3 hours after use of product.
  HRV refers to variation in the intervals between consecutive heart beats. Low HRV predicts poor prognosis and increased mortality in patients with cardiovascular disease and in apparently healthy subjects

OTHER OUTCOMES:
Clot strength and plasma levels of interleukin-6 (IL-6) and 8-isoprostane | up to 3 hours after use of product.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ganz, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Information might be disclosed as part of study activities to the FDA